CLINICAL TRIAL: NCT04365361
Title: Exploring the Psychological Impact of the COVID-19 on Higher Education Students
Brief Title: The Psychological Impact of the COVID-19 on Students.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Other Study IDs: UW20-298
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Mental Health Wellness 1
Keywords: Stress; Depression; Higher education students; Psychological impact
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 outbreak has been rapidly transmitted in late January 2020 and aroused enormous attention globally. The public at large may also experience boredom, disappointment, and irritability under the isolation measures. Depression and anxiety are common mental health problems experienced by university students. This survey aims to investigate the psychological impact of COVID 19 on students.

DETAILED DESCRIPTION:
The COVID-19 outbreak has been rapidly transmitted in late January 2020 and aroused enormous attention globally. Infected patients may develop severe and even fatal respiratory diseases (e.g., acute respiratory distress syndrome (ARDS) and acute respiratory failure) ending up in intensive care. Apart from physical suffering, it is not uncommon for confirmed or suspected cases of COVID-19 to suffer from great psychological pressure and other health-related problems. The limited knowledge of the COVID-19 and the overwhelming news may lead to anxiety and fear in the public. The public at large may also experience boredom, disappointment, and irritability under the isolation measures.

Depression and anxiety are common mental health problems experienced by university students. Being in higher education is associated with many stressors and transitional events, and students fall within the age range when common mental health problems are at their developmental peak. Depression and anxiety can impair students' academic performance and social functioning, cause significant burden at university, and potentially affect their future career opportunities. The study includes 2 parts. Part A is an online survey study with non-probabilistic convenience sampling and part B is focus group interviews.

This study aims to explore the psychological impact of COVID-19 and coping methods in higher education students.

ELIGIBILITY:
Inclusion Criteria:

• Higher education students aged 18 years and above

Exclusion Criteria:

• Subjects refuse to answer this questionnaire

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part A: An online survey study with non-probabilistic convenience sampling n=384
  Part B: Focus group interviews n=32
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress level | baseline
  measured by Stress Scale

SECONDARY OUTCOMES:
Anxiety and depressive symptoms | baseline
  measured by a 4-item Patient Health Questionnaire
Insomnia symptoms and the associated daytime impairment | baseline
  measured by 7-item Insomnia Severity Index
Psychological response to trauma | baseline
  measured by a 22-item Impact of Event Scale -Revised
Resilience | baseline
  measured by a 2-item Connor-Davidson Resilience Scale
Attitude and practice students regarding preventive measures | baseline
  measured by outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- LAI Agnes, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
It was not included in the participants' consent.

REFERENCES:
- [Background] Bao Y, Sun Y, Meng S, Shi J, Lu L. 2019-nCoV epidemic: address mental health care to empower society. Lancet. 2020 Feb 22;395(10224):e37-e38. doi: 10.1016/S0140-6736(20)30309-3. Epub 2020 Feb 7. No abstract available. PMID 32043982
- [Background] Hysenbegasi A, Hass SL, Rowland CR. The impact of depression on the academic productivity of university students. J Ment Health Policy Econ. 2005 Sep;8(3):145-51. PMID 16278502
- [Derived] Lai AYK, Cheung GOC, Choi ACM, Wang MP, Chan PSL, Lam AHY, Lo EWS, Lin CC, Lam TH. Mental Health, Support System, and Perceived Usefulness of Support in University Students in Hong Kong Amidst COVID-19 Pandemic: A Mixed-Method Survey. Int J Environ Res Public Health. 2022 Oct 9;19(19):12931. doi: 10.3390/ijerph191912931. PMID 36232227
- [Derived] Lai AY, Sit SM, Lam SK, Choi AC, Yiu DY, Lai TT, Ip MS, Lam TH. A Phenomenological Study on the Positive and Negative Experiences of Chinese International University Students From Hong Kong Studying in the U.K. and U.S. in the Early Stage of the COVID-19 Pandemic. Front Psychiatry. 2021 Dec 13;12:738474. doi: 10.3389/fpsyt.2021.738474. eCollection 2021. PMID 34966299